CLINICAL TRIAL: NCT01957202
Title: A Randomised, Double-blind, Placebo-controlled, 3 Way, Incomplete Block Cross Over Study in Subjects With Allergic Rhinitis to Assess the Effect of Once Daily Single and Repeat Doses of Intranasal Fluticasone Furoate/Levocabastine Fixed Dose Combination (FDC) Relative to Levocabastine and Fluticasone Furoate Alone on the Onset and Magnitude of Symptoms of Rhinitis in an Allergen Challenge Chamber
Brief Title: A Proof of Concept Study to Assess Effect of Fluticasone Furoate (FF)/Levocabastine Fixed Dose Combination (FDC) Compared With Levocabastine and FF Alone in Subjects With Allergic Rhinitis (AR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200286
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal
Keywords: levocabastine fixed dose combination, Rhinitis, Allergic, Perennial and Seasonal, Allergic Rhinitis, fluticasone furoate
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic | interventions — levocabastine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Each Subject will be assigned to a sequence of three treatments (e.g ABC, BCD, ACD): A=Two, 50 microliter (mcqL) sprays per nostril of FF, total dose 100 microgram (mcg); B=Two, 50 mcqL sprays per nostril of levocabastine, total dose 200 mcg; C=Two, 50 mcql sprays per nostril of FF/levocabastine FDC, total daily dose 100 mcg FF and 200 mcg levocabastine; D=Two, 50 mcql sprays per nostril of placebo. There will be a wash out period of 14-28 days between two treatment periods
  Interventions: Drug: FF/levocabastine; Drug: FF; Drug: levocabastine; Drug: Placebo

INTERVENTIONS:
Drug: FF/levocabastine — FF/levocabastine (25mcg/50 mcg) will be supplied as intranasal aqueous microsuspension in an amber glass bottle fitted with a white top actuated plastic metering atomising spray pump filled with a uniform white suspension. Two sprays in each nostril in the morning in a fasted state will be administered.
Drug: FF — FF (25mcg) will be supplied as intranasal aqueous microsuspension in an amber glass bottle fitted with a white top actuated plastic metering atomising spray pump filled with a uniform white suspension. Two sprays in each nostril in the morning in a fasted state will be administered.
Drug: levocabastine — levocabastine (50mcg) will be supplied as intranasal aqueous microsuspension in an amber glass bottle fitted with a white top actuated plastic metering atomising spray pump filled with a uniform white suspension. Two sprays in each nostril in the morning in a fasted state will be administered.
Drug: Placebo — Placebo will be supplied as intranasal aqueous microsuspension in an amber glass bottle fitted with a white top actuated plastic metering atomising spray pump filled with a uniform white suspension. Two sprays in each nostril in the morning in a fasted state will be administered.

SUMMARY:
This study will be a randomised, double blind, placebo controlled, 3-way, incomplete block crossover study to evaluate the effect of single and repeat doses of levocabastine, FF, placebo and a FDC of FF/levocabastine administration in AR subjects. The total expected study duration for each individual participating in the study will be a maximum of up to 20 weeks (including the screening and follow-up). This will be a three period study and subjects will be assigned to a sequence of three treatments. There will be a wash-out period of 14-28 days between two treatment periods. The rational for this study is to demonstrate proof of concept with the FDC of FF and levocabastine compared with each of the components administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AR, as determined by the presence of rhinitis symptoms that last for several months per year, for more than 1 year and are not attributed to infections or nasal abnormalities.
* Subjects have a TNSS score of >=6 during the screening allergen challenge chamber.
* Subjects have a positive skin prick test (wheal >=4 millimeter [mm]) for seasonal pollen at or within the 12 months preceding the screening visit.
* Subjects have a positive radioallergosorbent test (RAST) (>=class 2) for seasonal pollen at or within the 12 months preceding the screening visit.
* There are no conditions or factors that would make the subject unlikely to be able to stay in the chamber for 5 hours.
* Male/females between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination and laboratory tests. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kg and body mass index (BMI) within the range 19-30 kilogram per meter suare (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] >40 milli international unit per milliliter (MIU/milliliter [mL]) and estradiol <40 picogram per milliliter[pg/mL] (<147 picomole per liter [pmol/L]) is confirmatory).

Child-bearing potential with negative pregnancy test as determined by urine beta-human chorionic gonadotropin (β-hCG) test at screening or prior to dosing and;

* Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 1 week post-last dose
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subjects should be non-smokers, which for this study is defined as having smoked <10 packs per year in their lifetime, and have not smoked in the 6 months prior to the screening visit.
* alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT interval (QTc) values of triplicate electrocardiogram (ECGs) obtained over a brief recording period: Fridericia's QTC (QTcF) <450 milliseconds (msec).

Exclusion Criteria:

* Nasal abnormalities likely to affect the outcome of the study, that is nasal septal perforation, nasal polyps, sinusitis other nasal malformations.
* History of frequent nose bleeds
* Patients with rhinitis medicamentosa
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Significant renal impairment, which based on the opinion of the investigator, would preclude the subjects participation in the study.
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Murdoch RD, Bareille P, Ignar D, Miller SR, Gupta A, Boardley R, Zieglmayer P, Zieglmayer R, Lemel P, Horak F. The improved efficacy of a fixed-dose combination of fluticasone furoate and levocabastine relative to the individual components in the treatment of allergic rhinitis. Clin Exp Allergy. 2015 Aug;45(8):1346-55. doi: 10.1111/cea.12556. PMID 25900517
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 200286 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200286 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200286 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200286 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200286 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200286 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200286 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who met the eligibility criteria at Screening were randomized to 1 of 18 treatment sequences. The treatment phase was comprised of three 8-day treatment periods, each separated by a 14- to 28-day washout period.
Groups:
- Sequence 1: Levo 200 µg, FF 100 μg/Levo 200 μg, Placebo: Participants received levocabastine (Levo) 200 micrograms (µg), fluticasone furoate (FF) 100 μg/Levo 200 μg and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 μg once daily (OD) in the morning as 2 nasal spray (50 μg per spray) and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and placebo OD in the morning as 2 nasal sprays into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 2: Levo 200 µg, FF 100 μg, FF 100 μg/Levo 200 μg: Participants received Levo 200 µg, FF 100 µg and FF 100 μg/Levo 200 μg in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) and FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 3: Levo 200 µg, FF 100 μg/Levo 200 μg, FF 100 μg: Participants received Levo 200 µg, FF 100 μg/Levo 200 μg and FF 100 µg in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 4: Placebo, FF 100 μg, FF 100 μg/Levo 200 μg: Participants received placebo, FF 100 µg and FF 100 μg/Levo 200 μg in Treatment Periods 1, 2, and 3, respectively. Participants received the placebo OD in the morning as 2 nasal sprays and FF 100 µg OD in the morning as 2 nasal sprays and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 5: Placebo, FF 100 μg/Levo 200 μg, Levo 200 μg: Participants received placebo, FF 100 μg/Levo 200 μg and Levo 200 µg in Treatment Periods 1, 2, and 3, respectively. Participants received the placebo OD in the morning as 2 nasal sprays and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 6: FF 100 μg/Levo 200 μg, Placebo, Levo 200 μg: Participants received FF 100 μg/Levo 200 μg, placebo and Levo 200 µg in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and placebo OD in the morning as 2 nasal sprays and Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 7: FF 100 μg, Placebo 200 μg, FF 100 μg/Levo 200 μg: Participants received FF 100 µg, placebo and FF 100 μg/Levo 200 μg in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) and placebo OD in the morning as 2 nasal sprays and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 8: FF 100 μg/Levo 200 μg, FF 100 μg, Placebo: Participants received FF 100 μg/Levo 200 μg, FF 100 µg and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) and placebo OD in the morning as 2 nasal sprays into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 9: Placebo, FF 100 μg/Levo 200 μg, FF 100 μg: Participants received placebo, FF 100 μg/Levo 200 μg and FF 100 µg in Treatment Periods 1, 2, and 3, respectively. Participants received the placebo OD in the morning as 2 nasal sprays (50 μg per spray) and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 10: FF 100 μg, FF 100 μg/Levo 200 μg, Levo 200 μg: Participants received FF 100 µg, FF 100 μg/Levo 200 μg and Levo 200 µg in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 11: Levo 200 μg, Placebo, FF 100 μg/Levo 200 μg: Participants received Levo 200 µg, placebo and FF 100 μg/Levo 200 μg in Treatment Periods 1, 2, and 3, respectively. Participants received the Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) and placebo OD in the morning as 2 nasal sprays and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 12: FF 100 μg/Levo 200 μg, Levo 200 μg, FF 100 μg: Participants received FF 100 μg/Levo 200 μg, Levo 200 µg and FF 100 µg in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) and FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 13: FF 100 μg/Levo 200 μg, Levo 200 μg, Placebo: Participants received FF 100 μg/Levo 200 μg, Levo 200 µg and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) and placebo OD in the morning as 2 nasal sprays into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 14: FF 100 μg, FF 100 μg/Levo 200 μg, Placebo: Participants received FF 100 µg, FF 100 μg/Levo 200 μg and placebo in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and placebo OD in the morning as 2 nasal sprays into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 15: FF 100 μg/Levo 200 μg, FF 100 μg, Levo 200 μg: Participants received FF 100 μg/Levo 200 μg, FF 100 µg and Levo 200 µg in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) and Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 16: FF 100 μg/Levo 200 μg, Placebo, FF 100 μg: Participants received FF 100 μg/Levo 200 μg, placeboμg and FF 100 µg in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) and placebo µg OD in the morning as 2 nasal sprays and FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 17: FF 100 μg, Levo 200 μg, FF 100 μg/Levo 200 μg: Participants received FF 100 µg, Levo 200 µg and FF 100 μg/Levo 200 μg in Treatment Periods 1, 2, and 3, respectively. Participants received the FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) and Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
- Sequence 18: Placebo, Levo 200 μg, FF 100 μg/Levo 200 μg: Participants received placebo, Levo 200 µg and FF 100 μg/Levo 200 μg in Treatment Periods 1, 2, and 3, respectively. Participants received the placebo OD in the morning as 2 nasal sprays and Levo 200 μg OD in the morning as 2 nasal spray (50 μg per spray) and FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) into each nostril for 8 days. The three treatment periods were separated by a washout period of 14 to 28 days.
Period: Treatment Period 1 (8 Days)
Arm/Group | Sequence 1: Levo 200 µg, FF 100 μg/Levo 200 μg, Placebo | Sequence 2: Levo 200 µg, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 3: Levo 200 µg, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 4: Placebo, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 5: Placebo, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 6: FF 100 μg/Levo 200 μg, Placebo, Levo 200 μg | Sequence 7: FF 100 μg, Placebo 200 μg, FF 100 μg/Levo 200 μg | Sequence 8: FF 100 μg/Levo 200 μg, FF 100 μg, Placebo | Sequence 9: Placebo, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 10: FF 100 μg, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 11: Levo 200 μg, Placebo, FF 100 μg/Levo 200 μg | Sequence 12: FF 100 μg/Levo 200 μg, Levo 200 μg, FF 100 μg | Sequence 13: FF 100 μg/Levo 200 μg, Levo 200 μg, Placebo | Sequence 14: FF 100 μg, FF 100 μg/Levo 200 μg, Placebo | Sequence 15: FF 100 μg/Levo 200 μg, FF 100 μg, Levo 200 μg | Sequence 16: FF 100 μg/Levo 200 μg, Placebo, FF 100 μg | Sequence 17: FF 100 μg, Levo 200 μg, FF 100 μg/Levo 200 μg | Sequence 18: Placebo, Levo 200 μg, FF 100 μg/Levo 200 μg
Started | 3 | 6 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 6 | 3
Completed | 3 | 6 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 6 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (14 to 28 Days)
Arm/Group | Sequence 1: Levo 200 µg, FF 100 μg/Levo 200 μg, Placebo | Sequence 2: Levo 200 µg, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 3: Levo 200 µg, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 4: Placebo, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 5: Placebo, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 6: FF 100 μg/Levo 200 μg, Placebo, Levo 200 μg | Sequence 7: FF 100 μg, Placebo 200 μg, FF 100 μg/Levo 200 μg | Sequence 8: FF 100 μg/Levo 200 μg, FF 100 μg, Placebo | Sequence 9: Placebo, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 10: FF 100 μg, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 11: Levo 200 μg, Placebo, FF 100 μg/Levo 200 μg | Sequence 12: FF 100 μg/Levo 200 μg, Levo 200 μg, FF 100 μg | Sequence 13: FF 100 μg/Levo 200 μg, Levo 200 μg, Placebo | Sequence 14: FF 100 μg, FF 100 μg/Levo 200 μg, Placebo | Sequence 15: FF 100 μg/Levo 200 μg, FF 100 μg, Levo 200 μg | Sequence 16: FF 100 μg/Levo 200 μg, Placebo, FF 100 μg | Sequence 17: FF 100 μg, Levo 200 μg, FF 100 μg/Levo 200 μg | Sequence 18: Placebo, Levo 200 μg, FF 100 μg/Levo 200 μg
Started | 3 | 6 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 6 | 3
Completed | 3 | 6 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 6 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (8 Days)
Arm/Group | Sequence 1: Levo 200 µg, FF 100 μg/Levo 200 μg, Placebo | Sequence 2: Levo 200 µg, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 3: Levo 200 µg, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 4: Placebo, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 5: Placebo, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 6: FF 100 μg/Levo 200 μg, Placebo, Levo 200 μg | Sequence 7: FF 100 μg, Placebo 200 μg, FF 100 μg/Levo 200 μg | Sequence 8: FF 100 μg/Levo 200 μg, FF 100 μg, Placebo | Sequence 9: Placebo, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 10: FF 100 μg, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 11: Levo 200 μg, Placebo, FF 100 μg/Levo 200 μg | Sequence 12: FF 100 μg/Levo 200 μg, Levo 200 μg, FF 100 μg | Sequence 13: FF 100 μg/Levo 200 μg, Levo 200 μg, Placebo | Sequence 14: FF 100 μg, FF 100 μg/Levo 200 μg, Placebo | Sequence 15: FF 100 μg/Levo 200 μg, FF 100 μg, Levo 200 μg | Sequence 16: FF 100 μg/Levo 200 μg, Placebo, FF 100 μg | Sequence 17: FF 100 μg, Levo 200 μg, FF 100 μg/Levo 200 μg | Sequence 18: Placebo, Levo 200 μg, FF 100 μg/Levo 200 μg
Started | 3 | 6 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 6 | 3
Completed | 3 | 5 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 5 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout Period 2 (14 to 28 Days)
Arm/Group | Sequence 1: Levo 200 µg, FF 100 μg/Levo 200 μg, Placebo | Sequence 2: Levo 200 µg, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 3: Levo 200 µg, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 4: Placebo, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 5: Placebo, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 6: FF 100 μg/Levo 200 μg, Placebo, Levo 200 μg | Sequence 7: FF 100 μg, Placebo 200 μg, FF 100 μg/Levo 200 μg | Sequence 8: FF 100 μg/Levo 200 μg, FF 100 μg, Placebo | Sequence 9: Placebo, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 10: FF 100 μg, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 11: Levo 200 μg, Placebo, FF 100 μg/Levo 200 μg | Sequence 12: FF 100 μg/Levo 200 μg, Levo 200 μg, FF 100 μg | Sequence 13: FF 100 μg/Levo 200 μg, Levo 200 μg, Placebo | Sequence 14: FF 100 μg, FF 100 μg/Levo 200 μg, Placebo | Sequence 15: FF 100 μg/Levo 200 μg, FF 100 μg, Levo 200 μg | Sequence 16: FF 100 μg/Levo 200 μg, Placebo, FF 100 μg | Sequence 17: FF 100 μg, Levo 200 μg, FF 100 μg/Levo 200 μg | Sequence 18: Placebo, Levo 200 μg, FF 100 μg/Levo 200 μg
Started | 3 | 5 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 5 | 3
Completed | 3 | 5 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (8 Days)
Arm/Group | Sequence 1: Levo 200 µg, FF 100 μg/Levo 200 μg, Placebo | Sequence 2: Levo 200 µg, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 3: Levo 200 µg, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 4: Placebo, FF 100 μg, FF 100 μg/Levo 200 μg | Sequence 5: Placebo, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 6: FF 100 μg/Levo 200 μg, Placebo, Levo 200 μg | Sequence 7: FF 100 μg, Placebo 200 μg, FF 100 μg/Levo 200 μg | Sequence 8: FF 100 μg/Levo 200 μg, FF 100 μg, Placebo | Sequence 9: Placebo, FF 100 μg/Levo 200 μg, FF 100 μg | Sequence 10: FF 100 μg, FF 100 μg/Levo 200 μg, Levo 200 μg | Sequence 11: Levo 200 μg, Placebo, FF 100 μg/Levo 200 μg | Sequence 12: FF 100 μg/Levo 200 μg, Levo 200 μg, FF 100 μg | Sequence 13: FF 100 μg/Levo 200 μg, Levo 200 μg, Placebo | Sequence 14: FF 100 μg, FF 100 μg/Levo 200 μg, Placebo | Sequence 15: FF 100 μg/Levo 200 μg, FF 100 μg, Levo 200 μg | Sequence 16: FF 100 μg/Levo 200 μg, Placebo, FF 100 μg | Sequence 17: FF 100 μg, Levo 200 μg, FF 100 μg/Levo 200 μg | Sequence 18: Placebo, Levo 200 μg, FF 100 μg/Levo 200 μg
Started | 3 | 5 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 5 | 3
Completed | 3 | 5 | 6 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 3 | 6 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- FF 100 μg, Levo 200 μg, FF 100 μg/Levo 200 μg, Placebo: Participants received FF 100 µg, Levo 200 µg, FF 100 μg/Levo 200 μg and placebo once daily (OD) in the morning as 2 nasal sprays (FF: 25 µg per spray, Levo: 50 μg per spray, FF/Levo: 25 μg/50 μg per spray) into each nostril for 8 days each, in a crossover design. Treatment was given in one of 18 sequences in Periods 1, 2, and 3, (with a minimum of a 14-day washout period between treatments): BCD, BAC, BCA, DAC, DCB, CDB, ADC, CAD, DCA, ACB, BDC, CBA, CBD, ACD, CAB, CDA, ABC, DBC (A, FF 100 μg; B, Levo 200 μg; C, FF 100 μg/Levo 200 μg; D, placebo). On Day 1 and Day 8 of each treatment period, participants were subjected to an allergen challenge in a Vienna Challenge Chamber (VCC) for a 4-hour period, and the assessments were conducted 12-24 hours post-dose. All participants attended a follow-up visit of 14-28 days after their last dose, and the overall duration for participation in the study (screening to follow-up) was 20 weeks.
Arm/Group | FF 100 μg, Levo 200 μg, FF 100 μg/Levo 200 μg, Placebo
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.4 (8.91)
Gender [Count of Participants; unit: Participants]
  Female | 36
  Male | 35
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 2
  White - White/Caucasian/European Heritage | 69

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean of the Total Nasal Symptom Score (TNSS) (0-4) Hours (h) Post Start of Allergen Chamber Challenge on Day 8 of Each Treatment Period
Description: The TNSS (score of 0-12) is defined as the sum of the symptom scores for the four individual components (nasal congestion, rhinorrhea, nasal itch, and sneezing, each scored on 0-3 scale [0=none, 1=mild, 2=moderate, 3=severe]). TNSS was measured at the pre-allergen chamber challenge, and then every 15 minutes from 0 to 4 hours post start of the allergen chamber challenge. In the Environmental Exposure Chamber (EEC), aerosolized allergen was administered in a sealed chamber to evaluate the efficacy of antihistamines/other treatments. Weighted mean TNSS was calculated by dividing the value of the area under the response time curve over the 0-4 hours (calculated by trapezoidal rule) by the time interval of available data.
Time Frame: Day 8 of each treatment period (up to 80 days)
Population: Pharmacodynamic (PD) Population: all participants in the All Subjects Population (defined as all participants who received at least one dose of investigational product) and who also provided data from at least one PD assessment. Only those participants contributing data at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Placebo: Participants received placebo OD in the morning as 2 nasal sprays in each nostril for 8 days
- FF 100 μg: Participants received FF 100 µg OD in the morning as 2 nasal sprays (25 µg per spray) in each nostril for 8 days
- Levo 200 μg: Participants received Levo 200 µg OD in the morning as 2 nasal sprays (50 µg per spray) in each nostril for 8 days
- FF 100 μg/Levo 200 μg: Participants received FF 100 μg/Levo 200 µg OD in the morning as 2 nasal sprays (25 µg/50 μg per spray) in each nostril for 8 days
Arm/Group | Placebo | FF 100 μg | Levo 200 μg | FF 100 μg/Levo 200 μg
Number analyzed (Participants) | 34 | 54 | 53 | 66
Scores on a scale | 6.030 [5.350 to 6.710] | 4.189 [3.646 to 4.731] | 4.500 [3.955 to 5.044] | 1.933 [1.438 to 2.428]
Statistical Analysis 1: Comparison: FF 100 μg vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p < 0.0001, Mixed Model ANOVA; Mean Difference (Final Values) = -2.255, 95% CI 2-sided [-2.895 to -1.616]
Statistical Analysis 2: Comparison: Levo 200 μg vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p < 0.0001, Mixed Model ANOVA; Mean Difference (Final Values) = -2.566, 95% CI 2-sided [-3.208 to -1.925]
Statistical Analysis 3: Comparison: Placebo vs Levo 200 μg; Test type: Superiority or Other; p = 0.0003, Mixed Model ANOVA; Mean Difference (Final Values) = -1.531, 95% CI 2-sided [-2.342 to -0.719]
Statistical Analysis 4: Comparison: Placebo vs FF 100 μg; Test type: Superiority or Other; p < 0.0001, Mixed Model ANOVA; Mean Difference (Final Values) = -1.842, 95% CI 2-sided [-2.654 to -1.029]
Statistical Analysis 5: Comparison: Placebo vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p < 0.0001, Mixed Model ANOVA; Mean Difference (Final Values) = -4.097, 95% CI 2-sided [-4.857 to -3.337]
Statistical Analysis 6: Comparison: FF 100 μg vs Levo 200 μg; Test type: Superiority or Other; p = 0.3699, Mixed Model ANOVA; Mean Difference (Final Values) = -0.311, 95% CI 2-sided [-0.994 to 0.372]

2. Secondary Outcome: Weighted Mean of the Magnitude of Symptom Relief on Total Nasal Symptom Score (TNSS) (2-4) Hours (h) Post Start of Allergen Chamber Challenge on Day 1 of Each Treatment Period
Description: Magnitude of symptom relief was assessed by calculating change from pre-dose weighted mean TNSS (2-4h) post start of the allergen chamber challenge at Day 1. The pre-dose value was the maximum of the three pre-dose measurements (1h 15 minutes (min), 1h 30 min and 1h 45 min post start of the allergen chamber challenge). The TNSS (score of 0-12) is defined as the sum of the symptom scores for the four individual components (nasal congestion, rhinorrhea, nasal itch and sneezing, each scored on 0-3 scale [0=none, 1=mild, 2=moderate, 3=severe]).
Time Frame: Day 1 of each treatment period (up to 80 days)
Population: PD Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | FF 100 μg | Levo 200 μg | FF 100 μg/Levo 200 μg
Number analyzed (Participants) | 34 | 54 | 53 | 68
Scores on a scale | -1.335 [-1.861 to -0.810] | -0.904 [-1.332 to -0.476] | -2.588 [-3.018 to -2.157] | -2.267 [-2.658 to -1.877]
Statistical Analysis 1: Comparison: FF 100 μg vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p < 0.0001, Mixed Model ANOVA; Mean Difference (Final Values) = -1.364, 95% CI 2-sided [-1.853 to -0.874]
Statistical Analysis 2: Comparison: Levo 200 μg vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p = 0.1975, Mixed Model ANOVA; Mean Difference (Final Values) = 0.320, 95% CI 2-sided [-0.169 to 0.809]
Statistical Analysis 3: Comparison: Placebo vs Levo 200 μg; Test type: Superiority or Other; p < 0.0001, Mixed Model ANOVA; Mean Difference (Final Values) = -1.252, 95% CI 2-sided [-1.870 to -0.635]
Statistical Analysis 4: Comparison: Placebo vs FF 100 μg; Test type: Superiority or Other; p = 0.1648, Mixed Model ANOVA; Mean Difference (Final Values) = 0.432, 95% CI 2-sided [-0.179 to 1.042]
Statistical Analysis 5: Comparison: Placebo vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p = 0.0016, Mixed Model ANOVA; Mean Difference (Final Values) = -0.932, 95% CI 2-sided [-1.506 to -0.358]
Statistical Analysis 6: Comparison: FF 100 μg vs Levo 200 μg; Test type: Superiority or Other; p < 0.0001, Mixed Model ANOVA; Mean Difference (Final Values) = 1.684, 95% CI 2-sided [1.160 to 2.208]

3. Secondary Outcome: Weighted Mean of the Magnitude of Symptom Relief on Total Ocular Symptom Score (TOSS) (2-4) Hours (h) Post Start of Allergen Chamber Challenge on Day 1 of Each Treatment Period
Description: Magnitude of symptom relief was assessed by calculating change from pre-dose weighted mean TOSS (2-4h) post start of the allergen chamber challenge at Day 1. The pre-dose value was the maximum of the three pre-dose measurements (1h 15 minutes (min), 1h 30 min and 1h 45 min post start of the allergen chamber challenge). The TOSS (score of 0-9) is defined as the sum of the symptom scores for the three individual components (red, itchy, and tearing eyes, each scored on 0-3 scale [0=none, 1=mild, 2=moderate, 3=severe], average of two eyes).
Time Frame: Day 1 of each treatment period (up to 80 days)
Population: PD Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | FF 100 μg | Levo 200 μg | FF 100 μg/Levo 200 μg
Number analyzed (Participants) | 34 | 54 | 53 | 68
Scores on a scale | -0.097 [-0.431 to 0.237] | -0.272 [-0.537 to -0.007] | -0.633 [-0.901 to -0.365] | -0.446 [-0.683 to -0.209]
Statistical Analysis 1: Comparison: FF 100 μg vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p = 0.3052, Mixed Model ANOVA; Mean Difference (Final Values) = -0.174, 95% CI 2-sided [-0.508 to 0.160]
Statistical Analysis 2: Comparison: Levo 200 μg vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p = 0.2725, Mixed Model ANOVA; Mean Difference (Final Values) = 0.187, 95% CI 2-sided [-0.149 to 0.523]
Statistical Analysis 3: Comparison: Placebo vs Levo 200 μg; Test type: Superiority or Other; p = 0.0118, Mixed Model ANOVA; Mean Difference (Final Values) = -0.536, 95% CI 2-sided [-0.952 to -0.120]
Statistical Analysis 4: Comparison: Placebo vs FF 100 μg; Test type: Superiority or Other; p = 0.4049, Mixed Model ANOVA; Mean Difference (Final Values) = -0.175, 95% CI 2-sided [-0.588 to 0.239]
Statistical Analysis 5: Comparison: Placebo vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p = 0.0793, Mixed Model ANOVA; Mean Difference (Final Values) = -0.349, 95% CI 2-sided [-0.739 to 0.041]
Statistical Analysis 6: Comparison: FF 100 μg vs Levo 200 μg; Test type: Superiority or Other; p = 0.0478, Mixed Model ANOVA; Mean Difference (Final Values) = 0.361, 95% CI 2-sided [0.004 to 0.719]

4. Secondary Outcome: Weighted Mean of the Total Ocular Symptom Score (TOSS) (0-4) Hours (h) Post Start of Allergen Chamber Challenge on Day 8 of Each Treatment Period
Description: The TOSS (score of 0-9) is defined as the sum of the symptom scores for the three individual components (red, itchy, and tearing eyes , each scored on 0-3 scale [0=none, 1=mild, 2=moderate, 3=severe], average of two eyes). TOSS was measured at the pre-allergen chamber challenge, and then every 15 minutes from 0 to 4 hours post start of the allergen chamber challenge. In the Environmental Exposure Chamber (EEC), aerosolized allergen was administered in a sealed chamber to evaluate the efficacy of antihistamines/other treatments. Weighted mean TOSS was calculated by dividing the value of the area under the response time curve over the 0-4 hours (calculated by trapezoidal rule) by the time interval of available data.
Time Frame: Day 8 of each treatment period (up to 80 days)
Population: PD Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | FF 100 μg | Levo 200 μg | FF 100 μg/Levo 200 μg
Number analyzed (Participants) | 34 | 54 | 53 | 66
Scores on a scale | 1.321 [0.970 to 1.673] | 0.761 [0.465 to 1.057] | 0.621 [0.323 to 0.919] | 0.546 [0.268 to 0.824]
Statistical Analysis 1: Comparison: FF 100 μg vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p = 0.1502, Mixed Model ANOVA; Mean Difference (Final Values) = -0.215, 95% CI 2-sided [-0.509 to 0.079]
Statistical Analysis 2: Comparison: Levo 200 μg vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p = 0.6177, Mixed Model ANOVA; Mean Difference (Final Values) = -0.075, 95% CI 2-sided [-0.370 to 0.221]
Statistical Analysis 3: Comparison: Placebo vs Levo 200 μg; Test type: Superiority or Other; p = 0.0004, Mixed Model ANOVA; Mean Difference (Final Values) = -0.701, 95% CI 2-sided [-1.080 to -0.322]
Statistical Analysis 4: Comparison: Placebo vs FF 100 μg; Test type: Superiority or Other; p = 0.0035, Mixed Model ANOVA; Mean Difference (Final Values) = -0.560, 95% CI 2-sided [-0.934 to -0.187]
Statistical Analysis 5: Comparison: Placebo vs FF 100 μg/Levo 200 μg; Test type: Superiority or Other; p < 0.0001, Mixed Model ANOVA; Mean Difference (Final Values) = -0.775, 95% CI 2-sided [-1.123 to -0.428]
Statistical Analysis 6: Comparison: FF 100 μg vs Levo 200 μg; Test type: Superiority or Other; p = 0.3807, Mixed Model ANOVA; Mean Difference (Final Values) = 0.140, 95% CI 2-sided [-0.175 to 0.456]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment until the follow-up contact (up to 20 study weeks).
Description: SAEs and non-serious AEs were collected in members of the All Subject Population, comprised of all all participants who receive at least one dose of Investigational product.
Arm/Group | Placebo | FF 100 μg | Levo 200 μg | FF 100 μg/Levo 200 μg
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/54 | 0/53 | 0/68
Other Adverse Events (participants affected / at risk) | 2/34 | 1/54 | 1/53 | 3/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | FF 100 μg (N=54) | Levo 200 μg (N=53) | FF 100 μg/Levo 200 μg (N=68)
Headache (Nervous system disorders) | 2 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.